CLINICAL TRIAL: NCT06321302
Title: CRIMSON: A Multicentre, Randomised, Sham-controlled (and Active Controlled in the USA), Double-masked, 72-week Trial to Study the Safety, Tolerability, Pharmacokinetics, and Efficacy of 3 Dosing Regimens of Intravitreal BI 764524 in Patients With Moderately Severe to Severe Non-proliferative Diabetic Retinopathy
Brief Title: A Study to Test Whether BI 764524 Helps People With an Eye Condition Called Diabetic Retinopathy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1436-0007; 2023-508891-12-00 (Registry Identifier: CTIS); U1111-1299-0915 (Registry Identifier: Universal Trial Number)
Record Dates: First submitted 2024-03-14; First posted 2024-03-20 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BI 764524 (Experimental): BI 764524
  Interventions: Drug: BI 764524
- Sham comparator to BI 764524 (Sham Comparator): Sham comparator to BI 764524
  Interventions: Drug: Sham comparator to BI 764524
- Aflibercept (Eylea®) - US only (Active Comparator): Aflibercept (Eylea®) - US only
  Interventions: Drug: Aflibercept (Eylea®) - US only

INTERVENTIONS:
Drug: BI 764524 — BI 764524
  Arms: BI 764524
Drug: Sham comparator to BI 764524 — Sham comparator to BI 764524
  Arms: Sham comparator to BI 764524
Drug: Aflibercept (Eylea®) - US only — Aflibercept (Eylea®) - US only
  Arms: Aflibercept (Eylea®) - US only

SUMMARY:
This study is open to adults with diabetic retinopathy. People who have non-proliferative diabetic retinopathy of moderate or high severity can join the study.

The purpose of this study is to find out whether a medicine called BI 764524 helps people with diabetic retinopathy. The study also aims to find a suitable treatment plan for BI 764524. Participants are put into 5 groups by chance. Participants in groups 1, 2, and 3 get BI 764524. Over 1 year, they get a different number of injections of the same dose of BI 764524 injected into 1 eye. During some visits, participants may get a sham control, which is done like an eye injection but without a needle, so that participants will not know how many injections of BI 764524 they received. Participants in group 4 only get a sham control. Participants in group 5 (only in the USA) get aflibercept or sham injections during some visits. Aflibercept is a medicine already used to treat diabetic retinopathy.

Participants are in the study for one and a half years. During this time, they visit the study site at least 16 times. During this time, doctors regularly do eye exams and visual tests to assess the severity of participants' eye condition. After 1 year of treatment, researchers look at the number of participants with eye improvements. To do so, they compare eye damage and certain severe eye problems between the groups of participants. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
General inclusion criteria

* Diagnosis of diabetes mellitus (DM) under regular treatment with Haemoglobin A1c (HbA1c) (glycated haemoglobin) (HbA1c) <12%; DM should be under regular investigation by a trained specialist as per local standard of care prior to and during the trial
* Age ≥18 years at time of signing Informed Consent Form (ICF)

Ocular inclusion criteria: study eye

* Moderately severe to severe non-proliferative diabetic retinopathy (NPDR) (Diabetic Retinopathy Severity Scale (DRSS) 47 to 53) based on early treatment diabetic retinopathy study (ETDRS) 7-field grading as confirmed by the central reading centre (CRC) at screening
* Ultra-widefield fluorescein angiography (UWF-FA) image gradable for presence of retinal non-perfusion (RNP) as confirmed by the CRC at screening
* Visual acuity: best corrected visual acuity (BCVA) letter score of ≥49 letters (approximate Snellen equivalent of 20/100 or better) using ETDRS chart at starting distance of 4 meter (m) at screening
* Sufficiently clear ocular media, adequate pupillary dilation, and fixation to permit quality fundus imaging

Main exclusion criteria in study eye:

- Evidence of active retinal neovascularisation (NV) on clinical exam and/or ultra-widefield colour fundus photography (UWF-CFP) within the ETDRS 7-field, confirmed by the CRC grading

The following are permitted if, based on the assessment of the investigator, do not require acute treatment:

* Small neovascular lesions within the ETDRS 7-field that are detected only on UWF-FA, but not on clinical exam or colour fundus photography (CFP)
* Neovascularisations outside of the ETDRS 7-field on ultra-widefield imaging

  * Evidence of active NV of the iris (small iris tufts are not an exclusion) or in the anterior chamber angle
  * Prior pan-retinal photocoagulation (PRP). Peripheral scatter or targeted laser treatment in up to 1 quadrant outside the ETDRS 7-field area is permitted if it was performed at least 6 months prior to Day 1
  * CI-DME, defined as central subfield thickness (CST) ≥320 micrometer (μm) as measured by Heidelberg Spectralis optical coherence tomography (OCT) and confirmed by central reading centre (CRC) at screening (equivalent measurements from other OCT machines may be accepted); participants with a CST of 320-330 μm can be included if, in the opinion of the investigator, the participant is not expected to require treatment for CI-DME during the duration of the study (e.g. no profound impact on BCVA, stable CST, etc.)
  * Previous treatment in the study eye for NPDR and/or diabetic macular edema (DME) with intravitreal (IVT) anti-vascular endothelial growth factor (VEGF) (including anti-VEGF/Ang2) or short acting corticosteroid drugs (e.g. triamcinolone) within 6 months prior to Day 1 or dexamethasone intravitreal drug delivery system (Ozurdex) within 12 months prior to Day 1 (referred to elsewhere as 'previous IVT treatment').
  * Any previous IVT treatment other than anti-VEGF, and steroids. Previous fluocinolone acetonide intravitreal implant (Iluvien) is not allowed
  * Refractive error of more than -8 dioptres of myopia (spherical equivalent) in the study eye. For patients having undergone refractive or cataract surgery in the study eye, either the pre-operative refractive error or the axial length measurement should be used, at the investigator's discretion. Axial length should be less than 26 mm
  * Any concurrent or past ocular condition in the study eye which, in the judgement of the investigator, could:
* Require medical or surgical intervention during the study period to prevent or treat vision loss (e.g. advanced cataract, history of retinal detachment or macular hole (Stage 3 or 4) in the study eye)
* Could likely contribute to a significant loss of BCVA during the study period if left untreated (e.g. advanced epiretinal membrane and/or vitreomacular traction, active or history of optic neuritis in either eye)
* Contraindicate the use of the investigational drug, or may render the patient at high risk for treatment complications (e.g. active infectious or non-infectious conjunctivitis/keratitis in either eye; history of recurrent infectious or inflammatory ocular disease in either eye (e.g. uveitis)
* May affect interpretation of the study results (e.g. central atrophy of the retinal pigment epithelium or photoreceptors; age-related macular degeneration, hereditary retinal degenerative diseases, myopic macular degeneration, past, current or planned use of medications known to be toxic to the retina, lens or optic nerve (e.g. deferoxamine, chloroquine/hydroxychloroquine, chlorpromazine, phenothiazines, tamoxifen, nicotinic acid, and ethambutol); history of central serous chorioretinopathy, ischemic optic neuropathy or retinal vascular occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-09-17 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a ≥2-step improvement compared with baseline in Diabetic Retinopathy Severity Scale (DRSS) level in the study eye at Week 52 | At baseline and at Week 52
  The DRSS is a scale which can take on the following discrete values: 10, 20, 35, 43, 47, 53, 61, 65, 71, 75, 81, 85.
  Here 10 means "No retinopathy" and 85 means "Advanced proliferative diabetic retinopathy, with posterior fundus obscured, or centre of macula detached".
  Thus, a higher score means symptoms get worse.

SECONDARY OUTCOMES:
Occurrence of vision threatening complications (VTC)s in the study eye between baseline and Week 52 | At baseline and at Week 52
Absolute change from baseline of best corrected visual acuity (BCVA) [early treatment diabetic retinopathy study (ETDRS) letters] in the study eye at Week 52 | At baseline and at Week 52
  The BCVA score is the number of letters read correctly by the patient.
Absolute change from baseline of central subfield thickness (CST) [μm], as assessed by spectral domain optical coherence tomography (SD-OCT), in the study eye at Week 52 | At baseline and at Week 52
  μm= micrometer
Occurrence of a ≥2-step worsening of Diabetic Retinopathy Severity Scale (DRSS) in the study eye between baseline and Week 52 | At baseline and at Week 52
  The DRSS is a scale which can take on the following discrete values: 10, 20, 35, 43, 47, 53, 61, 65, 71, 75, 81, 85.
  Here 10 means "No retinopathy" and 85 means "Advanced proliferative diabetic retinopathy, with posterior fundus obscured, or centre of macula detached".
  Thus, a higher score means symptoms get worse.
Occurrence of proliferative diabetic retinopathy (PDR) and/or anterior segment neovascularisation (NV) in the study eye between baseline and Week 52 | At baseline and at Week 52
Development of centre-involved diabetic macular edema (CI-DME) in the study eye between baseline and Week 52 | At baseline and at Week 52
Occurrence of drug-related adverse events (AEs) between baseline and end of study (EOS) | up to 72 weeks
Occurrence of ocular AEs in the study eye between baseline and EOS | up to 72 weeks
Occurrence of ocular AEs of special interest in the study eye between baseline and EOS | up to 72 weeks

CONTACTS AND LOCATIONS:
Locations (88):
- United States (39):
  - Associated Retina Consultants, Ltd., Phoenix, Arizona
  - California Retina Consultants-Bakersfield-65523, Bakersfield, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retinal Diagnostic Center, Campbell, California
  - The Retina Partners, Encino, California
  - Lugene Eye Institute, Glendale, California
  - Retina Associates of Southern California, Huntington Beach, California
  - Byers Eye Institute, Palo Alto, California
  - California Eye Specialists Medical Group Inc, Pasadena, California
  - Retinal Consultants Medical Group, Sacramento, California
  - California Retina Consultants-Santa Maria-65510, Santa Maria, California
  - Bay Area Retina Associates - Walnut Creek, Walnut Creek, California
  - Colorado Retina Associates, Lakewood, Colorado
  - Retina Group of New England, PC, Waterford, Connecticut
  - Florida Retina Institute, Jacksonville, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Retina Consultants Of Hawaii, ‘Aiea, Hawaii
  - Maine Eye Center, Portland, Maine
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Deep Blue Retina Clinical Research PLLC, Southaven, Mississippi
  - NJRetina, Teaneck, New Jersey
  - Long Island Vitreoretinal Consultants, Great Neck, New York
  - Retina Vitreous Surgeons of Central NY, PC, Liverpool, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - EyeHealth Northwest, Portland, Oregon
  - Charleston Neuroscience Institute - Ladson, Ladson, South Carolina
  - Tennessee Retina, Nashville, Tennessee
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, PLLC, Austin, Texas
  - Austin Clinical Research, LLC, Austin, Texas
  - Retina Consultants of Texas, Katy, Texas
  - Valley Retina Institute, PA, McAllen, Texas
  - Austin Retina Associates, Round Rock, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Consultants of Texas, San Antonio, Texas
  - Retina Consultants of Texas - Schertz, Schertz, Texas
  - Retina Associates of Utah, Salt Lake City, Utah
- Germany (5):
  - Universitätsklinikum Bonn AöR, Bonn
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Dietrich-Bonhoeffer-Klinikum, Neubrandenburg
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
- Hungary (6):
  - Semmelweis University, Budapest
  - Budapest Retina Associations Kft., Budapest
  - Jahn Ferenc Del-Pest Hospital, Budapest
  - University Debrecen Hospital, Debrecen
  - Nozologen Kft., Pécs
  - Zala Megyei Szent Rafael Korhaz, Zala
- Italy (7):
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Fondazione IRCCS Ca'Granda-Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele S.r.l., Milan
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - IRCCS Fondazione Bietti, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Ospedali Riuniti di Ancona, Torrette Di Ancona
- Japan (14):
  - Akita University Hospital, Akita
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki-shi
  - Hayashi Eye Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Tokyo Medical University Hachioji Medical Center, Hachioji-shi
  - Kagawa University Hospital, Kagawa, Kita-gun
  - Kagoshima University Hospital, Kagoshima
  - Nara Medical University Hospital, Kashihara
  - Kobe University Hospital, Kobe
  - Shinshu University Hospital, Matsumoto-shi
  - National Hospital Organization Tokyo Medical Center, Meguro-ku
  - Aichi Medical University Hospital, Nagakute
  - Hyogo College of Medicine Hospital, Nishinomiya
  - Juntendo University Hospital, Tokyo
- Poland (5):
  - Klinika Okulistyczna, Bydgoszcz
  - Centrum Diagnostyki i Mikrochirurgii Oka-Lens Sp. z o.o., Olsztyn
  - Warsaw Ophthalmology Hospital, Warsaw
  - Centrum Medyczne Piasta 47 sp. z o.o., Wałbrzych
  - 4. Military Clinical Hospital with Polyclinic SP ZOZ, Wroclaw
- Emanuelli Research & Development Center, Arecibo, Puerto Rico
- Spain (5):
  - Hospital Universitari de Bellvitge, Barcelon
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari General de Catalunya, Sant Cugat Del Vallés
  - Hospital General Universitario de Valencia, Valencia
- United Kingdom (6):
  - East Suffolk and North Essex NHS Foundation Trust, Colchester
  - Royal Liverpool University Hospital, Liverpool
  - Moorfields Eye Hospital, London
  - Western Eye Hospital, London
  - King's College Hospital, London
  - Royal Victoria Infirmary, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents -upon signing of a 'Document Sharing Agreement'.For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com